CLINICAL TRIAL: NCT06759818
Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation on Postoperative Myocardial Injury in Elderly Patients Undergoing Thoracoscopic Surgery: a Prospective, Randomized Controlled Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Jiaxing University (Other)
Responsible Party: Principal Investigator, Qing-he Zhou, Affiliated Hospital of Jiaxing University, Affiliated Hospital of Jiaxing University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-LY-747
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-12

CONDITIONS: Myocardial Injury
Keywords: taVNS; myocardial injury; hs-cTnT; thoracoscopic surgery

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- transcutaneous vagus nerve stimulation (Experimental): ①The first adjustment requires electrical stimulation to break through the skin barrier. The first intervention is the day before the operation. The initial electrical stimulation frequency is 30Hz and the pulse width is 300μs. The frequency and pulse width are adjusted according to the individual feelings of the subject until they are tolerated by the subject. Maximum current stimulation without discomfort and lasting for 30 minutes; ② second time For the intervention, the subject is connected to the monitor after entering the surgery room. After observing that the subject's vital signs are within the normal range, the same stimulation frequency as the first time is immediately given for 30 minutes; ③ The third intervention is after the subject's surgery is completed. The same stimulation frequency was given in the resuscitation room until the patient was extubated and resuscitated.
  Interventions: Device: transcutaneous vagus nerve stimulation
- Sham stimulation group (Placebo Comparator): ① The first intervention is also the day before the operation. The frequency and pulse width are adjusted three times without turning on the machine, and the subject is asked if they have any feelings. After adjusting the frequency three times, no operation is performed for 30 minutes; ② The second intervention For the first intervention, after the monitor is connected in the operating room, the frequency and pulse width are not set, and it lasts for 30 minutes before being taken out; ③ For the third intervention, after the subject's surgery, earplugs are inserted in the recovery room, and the frequency and pulse width are not set. Remove the earplugs after extubation resuscitation is completed.
  Interventions: Device: Sham stimulation group

INTERVENTIONS:
Device: transcutaneous vagus nerve stimulation — ①The first adjustment requires electrical stimulation to break through the skin barrier. The first intervention is the day before the operation. The initial electrical stimulation frequency is 30Hz and the pulse width is 300μs. The frequency and pulse width are adjusted according to the individual feelings of the subject until they are tolerated by the subject. Maximum current stimulation without discomfort and lasting for 30 minutes; ② second time For the intervention, the subject is connected to the monitor after entering the surgery room. After observing that the subject's vital signs are within the normal range, the same stimulation frequency as the first time is immediately given for 30 minutes; ③ The third intervention is after the subject's surgery is completed. The same stimulation frequency was given in the resuscitation room until the patient was extubated and resuscitated.
  Arms: transcutaneous vagus nerve stimulation
Device: Sham stimulation group — ① The first intervention is also the day before the operation. The frequency and pulse width are adjusted three times without turning on the machine, and the subject is asked if they have any feelings. After adjusting the frequency three times, no operation is performed for 30 minutes; ② The second intervention For the first intervention, after the monitor is connected in the operating room, the frequency and pulse width are not set, and it lasts for 30 minutes before being taken out; ③ For the third intervention, after the subject's surgery, earplugs are inserted in the recovery room, and the frequency and pulse width are not set. Remove the earplugs after extubation resuscitation is completed.
  Arms: Sham stimulation group

SUMMARY:
This research group plans to design a prospective, double-blind, randomized controlled study to explore the effect of taVNS on hs-cTnT in elderly patients undergoing thoracoscopic surgery, and to evaluate the effect on perioperative myocardial injury and postoperative analgesia during thoracoscopic surgery.

DETAILED DESCRIPTION:
A small number of studies based on transcutaneous auricular vagus nerve stimulation have shown that it has good therapeutic effects on patients with cardiovascular disease, and is simple to operate, with few complications and low risks. However, thoracic surgery is closer to the heart and has a higher incidence of perioperative myocardial injury. , and hs-cTnT has become a biomarker that predicts myocardial injury. This research group plans to design a prospective, double-blind, randomized controlled study to explore the effect of taVNS on hs-cTnT in elderly patients undergoing thoracoscopic surgery, and to evaluate the effect on perioperative myocardial injury and postoperative analgesia during thoracoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥60 years old
2. Inpatients scheduled to undergo elective thoracoscopic lobectomy, segmentectomy, or wedge resection
3. ASA score of Ⅰ-Ⅲ
4. Able to communicate with the researcher Communicate and cooperate with patients completing assessment scales.

Exclusion Criteria:

1. Patients with congenital heart disease, coronary heart disease, myocardial infarction, severe heart block or implanted cardiac pacemaker
2. Patients with neurological diseases such as cerebral infarction, cerebral hemorrhage or stroke
3. Patients with pain, damage, infection or unhealed ear trauma in the area near the external auricle
4. Patients with a history of severe mental illness, abuse of analgesia or addiction to psychiatric drugs
5. Patients with severe digestive system diseases
6. Patients and their families who refuse surgical anesthesia or are unable to cooperate in completing the questionnaire
7. Pregnant women.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
high-sensitivity troponin T | The first day after surgery
  Trained researchers will draw 3-5ml blood samples before surgery, on the first day after surgery, and on the third day after surgery and store them in vacuum blood collection tubes containing lithium heparin. They will be temporarily stored in a refrigerator at 2-8°C within 24 hours. Sent to laboratory for analysis. All blood samples were analyzed by staff who received professional training in detecting Hs-cTnT using the Roche cobas e411 electrochemiluminescence fully automatic immunoassay analyzer.

SECONDARY OUTCOMES:
Myocardial injury after surgery | 30 days after surgery
  The 30-day MINS follow-up after surgery includes whether the patient has symptoms of myocardial ischemia such as chest tightness, angina pectoris, myocardial infarction, etc. It is also recommended that the patient come to the hospital for review of electrocardiogram and hs-cTnT and other indicators. Combining the current manufacturer-defined abnormal thresholds and the latest MINS study recommendations, we define MINS diagnostic criteria as hs-cTnT levels exceeding 14 ng/L during noncardiac surgery or within 30 days after surgery, and are at least 1 higher than the preoperative hs-cTnT level
high-sensitivity troponin T | the third day after surgery
  Trained researchers will draw 3-5ml blood samples before surgery, on the first day after surgery, and on the third day after surgery and store them in vacuum blood collection tubes containing lithium heparin. They will be temporarily stored in a refrigerator at 2-8°C within 24 hours. Sent to laboratory for analysis. All blood samples were analyzed by staff who received professional training in detecting Hs-cTnT using the Roche cobas e411 electrochemiluminescence fully automatic immunoassay analyzer.
NRS score 24 hours after surgery. | The three day after surgery
  Evaluate patients' resting pain scores 24 hours after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghe Zhou, Principal Investigator — Jiaxing University Affiliated Hospital; Mingzi An, MD, Study Director — Jiaxing University Affiliated Hospital.
Locations (1):
- The First Hospital of Jiaxing, Jiaxing, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackland GL, Abbott TEF, Jones TF, Leuwer M, Pearse RM; VISION-UK Investigators; University College Hospital; Royal Liverpool University Hospital; Leeds Teaching Hospitals. Early elevation in plasma high-sensitivity troponin T and morbidity after elective noncardiac surgery: prospective multicentre observational cohort study. Br J Anaesth. 2020 May;124(5):535-543. doi: 10.1016/j.bja.2020.02.003. Epub 2020 Mar 5. PMID 32147104